CLINICAL TRIAL: NCT04399408
Title: Mobile, Self-Operated, Home Ultrasound in Pregnancy - Safety, Efficacy and Usability
Brief Title: Instinct™ Ultrasound Device Safety, Efficacy and Usability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseNmore (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0004-19-RMC
Record Dates: First submitted 2020-05-10; First posted 2020-05-22 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2020-05

CONDITIONS: Ultrasonography, Prenatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Device users
  Interventions: Device: Obstetrics Ultrasound (non invasive)

INTERVENTIONS:
Device: Obstetrics Ultrasound (non invasive) — Participants are instructed to preform 1-3 short (3 minuets) ultrasound scans a day according to pre-defined steps.

SUMMARY:
Mobile medical devices for self-patient-use, are a rapidly evolving component of telehealth. Study examines the feasibility of using the INSTINCT® device, a portable self-use ultrasound system attached to a commercial smartphone in remote pregnancy assessment. Study aims to evaluate its safety, efficacy and usability.

DETAILED DESCRIPTION:
Study includes women carrying a singleton fetus at 14 to 40 gestational weeks. Women with multiple gestations, non-viable fetus at recruitment and those with a major fetal anatomical malformation or genetic syndrome are excluded. Each participant receives the device for a self-use period of 7-14 days, instructed to preform 1-3 scans a day. Each participant completes a self-assessment questionnaire which aims to evaluate satisfactory and usability (user experience and satisfaction). Each scan will be evaluated for the possibility to properly view fetal heart activity, amniotic fluid volume, fetal tone, fetal body and breathing movements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.
* Pregnancy week - 14-40.
* Fetus - single, no known genetic or anatomic defects.
* Able to understand and give informed consent.

Exclusion Criteria:

* Multiple pregnancy.
* Known genetic or anatomic defect to the fetus.
* Inability to understand how to operate the device or give informed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Safety - Device related SAE's | Through study completion until all subject gave birth, an average of 1 year
  The device will be deemed safe if all SAE will be classified as not device related

SECONDARY OUTCOMES:
User experience level | Through study completion, an average of 1 year
  User experience will be defined positive if the mean value of all answers to user satisfaction related questions in the CRF is better or equal 3.5 out of 5. Questions will be graded by a visual analog scale with scores of 1 to 5 (1=very poor, 5=very high)
Usability rating | Through study completion, an average of 1 year
  Usability will be defined positive if the mean value of all answers to usability related questions in the CRF is better or equal 3.5 out of 5. Questions will be graded by a visual analog scale with scores of 1 to 5 (1=very poor, 5=very high)
Device Sensitivity level | Through study completion, an average of 1 year
  Medical data recorded by the device will be defined useful if:
  At least 70% of 3 out of 5 tested parameters (Fetal Heartbeat, Movements, Tone, Breathing and Amniotic fluids) were classified by professional evaluator as "could be estimated".
  In more than 90% of scans, professional evaluator will be able to define Fetal Viability (identification of at least one of the following parameters: Fetal Heartbeat, Movements, Tone and Breathing)

CONTACTS AND LOCATIONS:
Overall Officials: Eran Hadar, M.D., Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No